CLINICAL TRIAL: NCT03256227
Title: Improving Veteran Adherence to Treatment for PTSD Through Partnering With Families
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIR 15-322
Record Dates: First submitted 2017-08-09; First posted 2017-08-21 (Actual); Results first posted 2024-06-14 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-01

CONDITIONS: Posttraumatic Stress Disorder
Keywords: Posttraumatic Stress Disorder; family therapy; patient adherence; Prolonged Exposure Therapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Patient Compliance

STUDY DESIGN:
Intervention Model Description: effectiveness-implementation Hybrid 1, 2-arm, pragmatic randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: Assessors are blinded to treatment condition
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Family Supported Prolonged Exposure (Experimental): The investigators propose to bring a family member into early educational sessions of PE, one of the most researched and efficacious treatments for PTSD, to increase family support for PE adherence. Strategies for how to engage with families are drawn from existing evidence-based approaches, including Motivational Interviewing and Behavioral Couples Therapy.
  Interventions: Behavioral: Family Supported Prolonged Exposure
- Standard Prolonged Exposure (Active Comparator): Standard Prolonged Exposure for PTSD as delivered in routine VA care.
  Interventions: Behavioral: Standard Prolonged Exposure

INTERVENTIONS:
Behavioral: Family Supported Prolonged Exposure — The investigators propose to bring a family member into early educational sessions of PE, one of the most researched and efficacious treatments for PTSD, to increase family support for PE adherence. Strategies for how to engage with families are drawn from existing evidence-based approaches, including Motivational Interviewing and Behavioral Couples Therapy.
  Arms: Family Supported Prolonged Exposure
Behavioral: Standard Prolonged Exposure — Standard Prolonged Exposure for PTSD as delivered in routine VA care.
  Arms: Standard Prolonged Exposure

SUMMARY:
Evidence-based psychotherapies (EBP) for PTSD, such as Prolonged Exposure (PE), result in clinically significant symptom relief for many. Yet, adherence to this treatment (i.e., session attendance and homework compliance), which is vital to ensuring recovery, can be poor. This project will test the effectiveness of improving family support for PE as a tool to improve Veterans' PE adherence. Reducing rates of dropout from PE will positively impact Veterans' health and well-being and lower the cost of treating PTSD. Additionally, despite congressional legislation and national mandates within VA/DoD for family involvement in PTSD care, there remains no proven strategies for how to routinely include family in traditional individual (i.e., one-on-one) EBPs for PTSD. This proposal will provide the initial test of a model of family engagement that can be translated to other problems faced by Veterans, including suicide prevention, traumatic brain injury (TBI) rehabilitation, and pain management, contributing to a broader evolution towards evidence-based, family-inclusive care.

DETAILED DESCRIPTION:
Impacts. This study aims to improve Veterans' adherence to evidence-based treatment for PTSD, through increasing family support for treatment. Improving retention rates in evidence-based PTSD treatment will positively impact Veterans' health and well-being, lower the cost of treating PTSD, and decrease long-term demand for PTSD services. If effective, this approach could help resolve national calls for routine inclusion of family involvement in PTSD treatment. Once demonstrated for PTSD, these strategies could be utilized for other conditions and problems relevant to Veteran populations (e.g., suicide prevention, traumatic brain injury (TBI) rehabilitation) and stimulate shifts across practice and policy to better routine and evidence-based involvement of families in care.

Background. PTSD occurs in as many as 1 in 5 combat Veterans and is associated with a host of negative, long-term consequences to the individual, their families, and society at large. Evidence-based psychotherapies, such as Prolonged Exposure (PE), result in clinically significant symptom relief for many. Yet, adherence to these treatments (i.e., session attendance and homework compliance), which is vital to ensuring recovery, can be poor. Engaging families in Veterans' treatment may provide a powerful method for promoting EBP adherence. The investigators data indicate that 70% of Veterans express some interest in involving their family in their care for PTSD; yet, only 17% of providers have had any contact with Veterans' families. The objective of the proposed study is to evaluate the effectiveness of improving family support as a tool to improve Veterans' EBP adherence. This research agenda directly addresses two VA HSR&D priorities:

* innovative mental health care;
* improving the quality of life for Veterans and their caregivers. The work aligns with the VHA Blueprint for Excellence and Strategic Plan through meeting the unique needs of military-service disabled Veterans, providing a novel treatment approach, and emphasizing patient- and family-centered care.

Objectives/Aims. Aim 1: To improve Veterans' adherence to PE through engaging families in care.

H1: Veterans randomized to family supported PE will attend more sessions (H1a) and report greater homework compliance (H1b) than Veterans randomized to standard PE delivered in routine care.

Aim 2: To improve the clinical outcomes of Veterans receiving PE through engaging families in care.

H2: Family supported PE will be more effective than standard PE in reducing PTSD severity and comorbid problems (depression, quality of life, relationship functioning) from baseline to posttreatment.

Aim 3: To examine barriers/facilitators of implementing family support for PE. Exploratory Aim: To identify mechanisms underlying adherence differences between treatment conditions.

The investigators will explore if adherence differences are mediated by changes on key social influence variables (family perceptions of treatment credibility, family support for PE, and family symptom accommodation).

Methods. The investigators are proposing a practical randomized controlled trial to compare Veteran adherence, and to PE with and without family attendance at PE's educational sessions, with the ultimate goal to improve Veterans' clinical outcomes. For Aim 3, the investigators will use a concurrent process evaluation to identify potential implementation facilitators and barriers to family involvement in PE within VA. Participants will include Veterans with clinically significant symptoms of PTSD across three sites, plus a family member or friend of the Veteran. Aim 1 outcome variables include session attendance and homework compliance. Aim 2 outcomes include PTSD symptom severity, depression, quality of life, and relationship functioning, measured monthly over the course of treatment. Key social influences (Exploratory Aim) will be assessed through brief weekly self-reports.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female veterans at least 18 years old. Recruitment is limited to Veterans enrolled in VHA care.
2. Participant meets DSM-5 diagnostic criteria for PTSD or subthreshold PTSD. Consistent with recommendations, subthreshold PTSD will be defined as endorsement of criteria A (trauma), F (duration), and G (impairment), with at least one symptom from each of the remaining diagnostic criteria (Brancu et al., 2016).
3. Has an intimate partner, family member, or friend with whom they have contact with at least 3 times a week
4. Willing to allow this person to participate in the study.
5. Provides informed consent.
6. Speaks and reads English.

Exclusion Criteria:

1. Current suicidal or homicidal ideation with intent and/or plan.
2. Meets DSM-5 criteria for a manic of psychotic episode in the past 3 months.
3. Meets DSM-5 diagnostic criteria for a severe substance use disorder in the past 3 months. Of note, subjects can be abusing or dependent upon nicotine or marijuana and still be included in the study.
4. Moderate relationship violence between the identified support person and the Veteran, defined as one or more episodes of severe violence in the past year (e.g., punched, kicked, or beat up).
5. Support person screens positive for PTSD on a self-report instrument (PCL).
6. Having an ongoing medical condition that would interfere with ability to attend weekly treatment sessions.
7. Having any planned upcoming major medical procedures over the next several months that would interfere with ability to attend weekly treatment sessions.
8. Veteran and/or SP fails to complete baseline survey
9. Episode of mania/psychosis in past 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura A. Meis, PhD, Principal Investigator — Minneapolis VA Health Care System, Minneapolis, MN
Locations (3):
- United States (3):
  - Atlanta VA Medical and Rehab Center, Decatur, GA, Decatur, Georgia
  - VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan
  - Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Meis LA, Glynn SM, Spoont MR, Kehle-Forbes SM, Nelson D, Isenhart CE, Eftekhari A, Ackland PE, Linden EB, Orazem RJ, Cutting A, Hagel Campbell EM, Astin MC, Porter KE, Smith E, Chuick CD, Lamp KE, Vuper TC, Oakley TA, Khan LB, Keckeisen SK, Polusny MA. Can families help veterans get more from PTSD treatment? A randomized clinical trial examining Prolonged Exposure with and without family involvement. Trials. 2022 Mar 30;23(1):243. doi: 10.1186/s13063-022-06183-2. PMID 35354481

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Family Supported Prolonged Exposure | Standard Prolonged Exposure
Started | 64 | 64
Completed (Completed treatment therapy) | 36 | 25
Not Completed | 28 | 39

BASELINE CHARACTERISTICS:
Population: Includes baseline data for all Veteran participants in the study
Groups:
- Total: Total of all reporting groups
Arm/Group | Family Supported Prolonged Exposure | Standard Prolonged Exposure | Total
Number analyzed (Participants) | 64 | 64 | 128
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.30 (14.70) | 51.23 (15.04) | 50.38 (14.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 11 | 25
  Male | 50 | 53 | 103
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Black | 14 | 14 | 28
  Race/Ethnicity: Hispanic/Latino | 1 | 4 | 5
  Race/Ethnicity: White | 41 | 36 | 77
  Race/Ethnicity: Multiracial | 4 | 6 | 10
  Race/Ethnicity: Unknown | 4 | 4 | 8
Lives with Significant Other [Count of Participants; unit: Participants] | 48 | 40 | 88

OUTCOME MEASURES:

1. Primary Outcome: Session Attendance
Description: Number of treatment sessions attended by the participant
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: sessions
Arm/Group | Family Supported Prolonged Exposure | Standard Prolonged Exposure
Number analyzed (Participants) | 64 | 64
sessions | 6.77 (3.99) | 5.56 (4.16)

2. Secondary Outcome: PTSD Checklist for DSM-5 (PCL-5)
Description: The PCL-5 is a 20-item self-report measure that assesses the 20 DSM-5 symptoms of PTSD. Range of scale is 0-80 and can be obtained by summing the scores for each of the 20 items. Higher scores indicate higher PTSD symptom levels.
Time Frame: 16 weeks
Population: Veterans who completed PCL5 measure at post treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Family Supported Prolonged Exposure | Standard Prolonged Exposure
Number analyzed (Participants) | 62 | 62
score on a scale | 51.56 (12.60) | 53.79 (12.54)

ADVERSE EVENTS:
Time Frame: Treatment initiation through 3 month follow-up, up to 40 weeks.
Description: This is a minimal risk study, so likelihood of mortality is zero.
Arm/Group | Family Supported Prolonged Exposure | Standard Prolonged Exposure
All-Cause Mortality (participants affected / at risk) | 0/64 | 0/64
Serious Adverse Events (participants affected / at risk) | 2/64 | 2/64
Other Adverse Events (participants affected / at risk) | 17/64 | 20/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Family Supported Prolonged Exposure (N=64) | Standard Prolonged Exposure (N=64)
Severe Suicidal ideation (Psychiatric disorders) | 2 (2) | 1 (1)
Psychological decompisation (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Family Supported Prolonged Exposure (N=64) | Standard Prolonged Exposure (N=64)
ER visit (General disorders) | 11 (24) | 14 (18)
Hospitalization (General disorders) | 8 (14) | 6 (9)
Mild Suicidal ideation (Psychiatric disorders) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
Smaller number of subjects analyzed than originally proposed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-08): https://cdn.clinicaltrials.gov/large-docs/27/NCT03256227/Prot_SAP_000.pdf